CLINICAL TRIAL: NCT02081365
Title: Clinical Management of Anxiety and Access to Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4100054871
Record Dates: First submitted 2013-12-17; First posted 2014-03-07 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-12

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Anxiety Computerized Dental Anxiety Treatment (Experimental): Computer based CBT intervention before the scheduled dental appoinment (1.5 hours)
  Interventions: Behavioral: Computerized Dental Anxiety Treatment
- High Anxiety Wailist Control (No Intervention)

INTERVENTIONS:
Behavioral: Computerized Dental Anxiety Treatment — The Computerized Dental Anxiety Treatment Program consists of treatment modules that are be delivered through a computer. The modules use Cognitive Behavioral Therapy (CBT) to assist the participant in preparing a personal plan for managing his/her dental anxiety. The program incorporates a range of CBT techniques, including cognitive restructuring, exposure, and motivational interviewing.
  Arms: High Anxiety Computerized Dental Anxiety Treatment

SUMMARY:
Dental and health anxiety are common and potentially distressing problems, for both patients and health care providers. Anxiety has been identified as a barrier to regular dental visits and as an important target for enhancement of oral health-related quality of life. possible groups, (1) high dental anxiety and (2) low dental anxiety. The study aimed to develop and evaluate a computerized cognitive-behavioral therapy dental anxiety intervention (C-CBT) that could be easily implemented in dental healthcare settings.

A cognitive-behavioral protocol based on psychoeducation, exposure to feared dental procedures, and cognitive restructuring was developed. A randomized controlled trial was conducted (N=151) to test its efficacy. Consenting adult dental patients who met inclusion (e.g., high dental anxiety) and exclusion criteria were randomized to one of two groups, (1) immediate treatment (IT) (n=74) or (2) a waitlist control (WL) (n=77).

DETAILED DESCRIPTION:
Analyses of covariance (ANCOVAs) based on intention to treat analyses were used to compare the two groups on dental anxiety, fear, avoidance, and overall severity of dental phobia. Baseline scores on these outcomes were entered into the analyses as covariates.

ELIGIBILITY:
Inclusion Criteria:

* high dental anxiety
* fluent in spoken and written English

Exclusion Criteria:

* unable to provide written, informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marisol Tellez, Ph.D., Principal Investigator — Temple University Kornberg School or Dentistry
Locations (1):
- Temple University Kornberg School of Dentistry, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tellez M, Potter CM, Kinner DG, Jensen D, Waldron E, Heimberg RG, Myers Virtue S, Zhao H, Ismail AI. Computerized Tool to Manage Dental Anxiety: A Randomized Clinical Trial. J Dent Res. 2015 Sep;94(9 Suppl):174S-80S. doi: 10.1177/0022034515598134. Epub 2015 Jul 22. PMID 26202996

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Treatment: Before the intervention, participants completed self-report questionnaires and a telephone diagnostic interview. Participants in the immediate treatment group were asked to come in 1.5 hours before a previously scheduled dental appointment to complete the computerized cognitive-behavioral therapy dental anxiety intervention (C-CBT).
  The C-CBT consisted of a single-session, one-hour computerized intervention that assisted the participant in building skills for managing his or her dental anxiety.
  One month after the dental appointment, participants were contacted by phone and asked to complete follow-up assessments.
- Waiting List Control: Before their dental appointments, participants completed self-report questionnaires and a telephone diagnostic interview. Waiting list control participants attended their scheduled dental appointment without receiving the computerized cognitive-behavioral therapy dental anxiety intervention but were offered the opportunity to receive the same intervention following all of their study assessments.
  One month after the dental appointment, participants were contacted by phone and asked to complete follow-up assessments.
Period: Overall Study
Arm/Group | Immediate Treatment | Waiting List Control
Started | 74 | 77
Received Allocated Intervention | 46 | 59
Completed | 44 | 54
Not Completed | 30 | 23

BASELINE CHARACTERISTICS:
Population: Patients were between 18 and 70 years, fluent in English, had scheduled a dental treatment appointment at the clinic, were willing and able to give informed written consent, met criteria for high dental anxiety based on the Modified Dental Anxiety Scale, and endorsed at least some oral-health related impairment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment | Waiting List Control | Total
Number analyzed (Participants) | 74 | 77 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (12.8) | 44.6 (13.6) | 44.7 (13.1)
Gender [Count of Participants; unit: Participants]
  Female | 52 | 41 | 93
  Male | 22 | 36 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 53 | 58 | 111
  Unknown or Not Reported | 16 | 14 | 30
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 18 | 38
  Black or African American | 34 | 44 | 78
  Asian | 2 | 2 | 4
  Other | 6 | 3 | 9
  Not reported/missing | 12 | 10 | 22
MDAS Baseline Score [Mean (Standard Deviation); unit: units on a scale] — Modified Dental Anxiety Scale Baseline Score (0-25 scale). We considered patients who scored > 19 on the MDAS at baseline or endorsed at least two MDAS items > 4 to have high dental anxiety.
  units on a scale | 19.5 (2.9) | 19.6 (2.6) | 19.5 (2.8)
ADIS Specific Phobia Fear Rating [Mean (Standard Deviation); unit: units on a scale] — Anxiety Disorders Interview Schedule for DSM-IV Specific Phobia Module Fear Rating 0 (none) to 8 (very severe).
  units on a scale | 5.6 (1.3) | 5.2 (1.4) | 5.4 (1.3)
ADIS Specific Phobia Avoidance Rating [Mean (Standard Deviation); unit: units on a scale] — Anxiety Disorders Interview Schedule for DSM-IV Specific Phobia Module Avoidance Rating (0-8 scale). 0 (none) to 8 (very severe).
  units on a scale | 4.6 (2.2) | 3.9 (2.5) | 4.2 (2.4)
ADIS Specific Phobia Clinical Severity Rating [Mean (Standard Deviation); unit: units on a scale] — Anxiety Disorders Interview Schedule for DSM-IV Specific Phobia Module Clinical Severity Rating (0-8 scale) 0 (none) to 8 (very severe); a CSR > 4 indicated that the participant met criteria for diagnosis of dental phobia.
  units on a scale | 5.3 (1.4) | 4.8 (1.6) | 5.0 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Modified Dental Anxiety Scale
Description: The Modified Dental Anxiety Scale a five-item self-report measure that assesses fear of dental procedures, including drilling, scaling and polishing (i.e., cleaning), and local anesthetic injections. Sample items include, "If you went to your dentist for treatment tomorrow, how would you feel?" and "If you were about to have your tooth drilled, how would you feel?" Items are rated on a five-point Likert-type scale ranging from 1 (not anxious) to 5 (extremely anxious). Scale 0-25. We considered patients who scored > 19 on the MDAS at baseline or endorsed at least two MDAS items > 4 to have high dental anxiety.
Time Frame: Change from one week before dentist appointment to 1 month after dentist appointment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Treatment | Waiting List Control
Number analyzed (Participants) | 74 | 77
units on a scale
  Baseline | 19.5 (0.34) | 19.6 (0.30)
  One month follow up | 15.4 (0.74) | 17.6 (0.63)
Statistical Analysis 1: Comparison: Immediate Treatment vs Waiting List Control; Comparison of two groups at 1 month follow up with baseline value as the covariate; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 2.2, 95% CI 2-sided [.74 to 3.55]

2. Secondary Outcome: Change in Clinical Severity Rating for Specific Phobia Module of Anxiety Disorders Interview Schedule for DSM-IV
Description: The Anxiety Disorders Interview Schedule for DSM-IV is a semi-structured diagnostic interview for assessing DSM-IV criteria for current anxiety, depressive, somatoform, and substance use disorders. For the present investigation, only the specific phobia module of the ADIS-IV was administered to assess the presence and severity of a current diagnosis of dental phobia. Various aspects of dental phobia were assessed using the specific phobia module of the ADIS-IV. Interviewers assessed participants' anxiety and avoidance of dental procedures on scales that ranged from 0 (none) to 8 (very severe). They also rated patients' overall distress and impairment due to their dental phobia symptoms and assigned a clinician's severity rating (CSR) that also ranged from 0 (none) to 8 (very severe); a CSR > 4 indicated that the participant met criteria for diagnosis of dental phobia.
Time Frame: Change from one week before dental appointment to one-month after dental appointment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Treatment | Waiting List Control
Number analyzed (Participants) | 52 | 63
units on a scale
  Baseline | 5.3 (0.19) | 4.8 (0.20)
  One month follow up | 3.4 (0.27) | 4.0 (0.23)
Statistical Analysis 1: Comparison: Immediate Treatment vs Waiting List Control; Comparison of two groups at 1 month follow up with baseline value as the covariate; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 0.98, 95% CI 2-sided [.39 to 1.57]

3. Secondary Outcome: Change in Fear Rating for Specific Phobia Module of Anxiety Disorders Interview Schedule for DSM-IV
Description: as for outcome 2
Time Frame: Change from one week before appointment to one month after appointment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Treatment | Waiting List Control
Number analyzed (Participants) | 52 | 63
units on a scale
  Baseline | 5.6 (0.17) | 5.2 (0.17)
  One month follow up | 3.8 (0.26) | 4.8 (0.23)
Statistical Analysis 1: Comparison: Immediate Treatment vs Waiting List Control; Comparison of two groups at 1 month follow up with baseline value as the covariate; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [.61 to 1.85]

4. Secondary Outcome: Change in Avoidance Rating for Specific Phobia Module of Anxiety Disorders Interview Schedule for DSM-IV
Description: as for outcome 2
Time Frame: Change from one week before appointment to one month after appointment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Immediate Treatment | Waiting List Control
Number analyzed (Participants) | 52 | 63
units on a scale
  Baseline | 4.6 (0.31) | 3.9 (0.32)
  One month follow up | 1.3 (0.31) | 1.0 (0.29)
Statistical Analysis 1: Comparison: Immediate Treatment vs Waiting List Control; Comparison of two groups at 1 month follow up with baseline value as the covariate; Test type: Superiority or Other; p < 0.05, ANCOVA; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [.01 to 1.64]

ADVERSE EVENTS:
Arm/Group | Immediate Treatment | Waiting List Control
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/77
Other Adverse Events (participants affected / at risk) | 0/74 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No